CLINICAL TRIAL: NCT02785094
Title: Education and Social Media Versus Non-Indicated Caesarean Section Rate in Egypt
Status: Completed | Type: Observational
Sponsor: Talkha Central Hospital (Other Government)
Responsible Party: Principal Investigator, Amro Mohamed Ibrahim Ibrahim Hetta, Dr. Amro M. Hetta, Talkha Central Hospital
Other Study IDs: OG3
Record Dates: First submitted 2016-05-23; First posted 2016-05-27 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Complications; Cesarean Section
Keywords: Caesarean Section Rate; Primigravida
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- A: Group of High Education level
  Interventions: Behavioral: Observation
- B: Group of Low/Non Education level
  Interventions: Behavioral: Observation
- C: Group has Accessibility to Social Media
  Interventions: Behavioral: Observation
- D: Group has not Accessibility to Social Media
  Interventions: Behavioral: Observation

INTERVENTIONS:
Behavioral: Observation — Observation of Participants' behaviour

SUMMARY:
This study focus on measuring effect of Egyptian Primigravidas' education level and accessibility to social media on rate of maternal request option offered for non-indicated primary caesarean section.

DETAILED DESCRIPTION:
A caesarean section (CS) is a life-saving surgical procedure when certain complications arise during pregnancy and labour. However, it is a major surgery and is associated with immediate maternal and perinatal risks and may have implications for future pregnancies as well as long-term effects that are still being investigated. The use of CS has increased dramatically worldwide in the last decades particularly in middle- and high-income countries, and some studies showing a link between increasing CS rates and poorer outcomes, and reasons for this increase are multifactorial and not well-understood.

In Egypt the CS rate according to WHO (World Health Organization),Health report (2010) is 27.6 %. Egypt also is considered to be the highest African country in CS rate (51.8 %), in which CS rate rose from 4.6 % to 51.8 % over the 24 year period (1990-2014), and more than half of all women give birth by CS in Egypt without much difference between urban and rural areas.

Slightly more than half of the live births in the five-year period before 2014 Egypt Demographic and Health survey were by CS, and 60 % of primigravidas delivered by CS.

Updated indications of primary CS including option of maternal request as one of these indications were reported in both RCOG (Royal College of Obstetricians and Gynaecologists) Press report (2001) and RCOG CS various guidelines.

Recently, the Egyptian public opinion deviated to obstetricians' desire for self financial benefits to be the major cause of increasing Egypt CS rates; depending on newspaper articles and social media talks.

ELIGIBILITY:
Inclusion Criteria:

* Full term with gestational age (G.A) more than or equal 39 weeks.
* Acceptance to answer study short questionnaire to determine eligible participants for each cohort.

Exclusion Criteria:

* Multiparity.
* History of previous Caesarean Section/s.
* Any Mental or Physical disabilities.
* Disapproval for answering a predefined short questionnaire related to study.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Primigravidas whom been carefully counselled, and the overall risks and benefits of caesarean section and vaginal birth, and IOL for prolonged pregnancy discussed with.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Actual)
Dates: Start 2016-06; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of Primigravidas who request a Non-Indicated CS | Up to 2 weeks
  Number of Primigravidas who request a Non-Indicated CS.

SECONDARY OUTCOMES:
Number of Primigravidas who refused to have a trial of IOL (Induction of Labour), as an index for deviated intention to request a Non-Indicated CS | Up to 24 hours
  Number of Primigravidas who refused to have a trial of IOL (Induction of Labour), as an index for deviated intention to request a Non-Indicated CS.

CONTACTS AND LOCATIONS:
Overall Officials: Amro M Hetta, M.B., Ch.B., Principal Investigator — Talkha Central Hospital
Locations (1):
- Talkha Central Hospital, Al Mansurah, Al-Dakahliya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Betran AP, Ye J, Moller AB, Zhang J, Gulmezoglu AM, Torloni MR. The Increasing Trend in Caesarean Section Rates: Global, Regional and National Estimates: 1990-2014. PLoS One. 2016 Feb 5;11(2):e0148343. doi: 10.1371/journal.pone.0148343. eCollection 2016. PMID 26849801
- [Background] Gibbons L, Belizán JM, Lauer JA, Betrán AP, Merialdi M, Althabe F. The global numbers and costs of additionally needed and unnecessary caesarean sections performed per year: overuse as a barrier to universal coverage. World health report 2010, 30: 1-31.
- [Background] Ministry of Health and Population [Egypt], El-Zanaty and Associates [Egypt], and ICF International. 2015. Egypt Demographic and Health Survey 2014. Cairo, Egypt and Rockville, Maryland, USA: Ministry of Health and Population and ICF International.
- [Background] Thomas J, Paranjothy S. Royal College of Obstetricians and Gynaecologists Clinical Effectiveness Support Unit. National Sentinel Caesarean Section Audit Report. London: RCOG press; 2001.